CLINICAL TRIAL: NCT05191719
Title: Neurotomy to Treat Synkinesis Following Peripheral Facial Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rebecka Ohm (Other)
Responsible Party: Sponsor-Investigator, Rebecka Ohm, Birgit Stark, MD, associate professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: K2018-5656
Record Dates: First submitted 2021-11-07; First posted 2022-01-13 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Facial Paralysis; Facial Palsy; Peripheral Facial Palsy; Peripheral Facial Paralysis; Bell Palsy; Synkinesis
MeSH Terms: conditions — Facial Paralysis; Bell Palsy; Synkinesis | interventions — Botulinum Toxins, Type A; Denervation

STUDY DESIGN:
Intervention Model Description: All study participants are evaluated with and without the effect Botox treatment before surgery. Botox is the gold standard treatment and used as a comparator. As all study patients have failed current evidence based treatment options, a comparative group not receiving treatment would imply a strong information bias.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botox (Active Comparator)
  Interventions: Procedure: Botox injection; Procedure: Neurotomy
- Neurotomy (Experimental)
  Interventions: Procedure: Botox injection; Procedure: Neurotomy

INTERVENTIONS:
Procedure: Botox injection — Comparator, current gold standard
Procedure: Neurotomy — Surgical procedure

SUMMARY:
The purpose of this study is to evaluate neurotomy as an alternative treatment to Botox injections for severe synkinesis following peripheral facial palsy

DETAILED DESCRIPTION:
Patients with severe synkinesis treated at Karolinska University Hospital with Botox injections with unsatisfying results are invited to participate in this study aiming to evaluate surgical neurotomy to synkinesis causing branches of the facial nerve.

Surgical procedure:

Small branches of the facial nerve are identified under microscopic magnification. Using a precise nerve stimulator the movement each nerve branch elicits is evaluated as normal or synkinetic. Pathological branches are then parted while normal functioning nerve branches are left intact.

Evaluation procedure:

Study participants are measured in a multimodal manner at 5 different time points during the study period; at study start, with and without Botox effect before surgery, and at 6 and 12 months after surgery. Evaluation methods:

* Clinical evaluation with Sunnybrook facial grading scale, blinded to observer from video recordings at the end of the study
* Neurophysiological measurements,
* Quality of life, measured with validated questionnaires FaCE, FDI, SAQ
* Reports of potential side effects, using Clavien-Dindo classification as well as free text

ELIGIBILITY:
Inclusion Criteria:

* Synkinesis following peripheral facial palsy
* Sunnybrook score <61
* Botox injections at least 3 times a year
* Have received at least 3 Botox injections
* Botox injections not satisfying treatment
* Read and signed written consent

Exclusion Criteria:

* Synkinesis since less than 2 years
* Contractures in facial muscles
* Other planned surgery in the face during study period
* Smoking
* Uncontrolled hypertension
* Diabetes mellitus
* Pregnancy or breast feeding
* Severe systemic disease (ASA 3-4)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Sunnybrook facial grading scale | Baseline, 4 months after Botox (no effect), 2-4 weeks after Botox (max effect), 6 and 12 months after surgery
  Improvement through less synkinesis and better voluntary movement

SECONDARY OUTCOMES:
Quality of life questionnaire | 4 months after Botox (no effect), 2-4 weeks after Botox (max effect), 6 and 12 months after surgery
  Facial Clinimetric Evaluation Scale (FaCE)
Quality of life questionnaire | 4 months after Botox (no effect), 2-4 weeks after Botox (max effect), 6 and 12 months after surgery
  Facial Disability Index (FDI)
Quality of life questionnaire | 4 months after Botox (no effect), 2-4 weeks after Botox (max effect), 6 and 12 months after surgery
  Synkinesis Assessment Questionnaire (SAQ)
Neurophysiological examination, electromyography (EMG). | 4 months after Botox (no effect), 2-4 weeks after Botox (max effect), just before surgery, 6 and 12 months after surgery
  Severity of synkinesis evaluation using EMG calculations (turns and root mean square (RMS)) compared to the healthy hemiface (reference).
Number of Botox injections | Baseline, 12 months after surgery
  Decrease to no future need
Side effects | Baseline, 2-4 weeks after Botox (max effect), 6 and 12 months after surgery
  Clavien-Dindo Classification
Side effects | Baseline, 2-4 weeks after Botox (max effect), 6 and 12 months after surgery
  Free text, in order to capture all possible side effects of treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Stark, MD, PhD, Principal Investigator — Karolinska Institute/Karolinska University Hospital
Locations (1):
- Karolinska University Hospital/Karolinska Institute, Stockholm, Sweden